CLINICAL TRIAL: NCT03712761
Title: Supplementation of a Leucine-Enriched Dairy Protein Blend: Effects on Plasma Amino Acids in Older Adults
Brief Title: Supplementation of a Leucine-Enriched Dairy Protein Blend
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Other Study IDs: 2502
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Dietary Protein Supplementation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Supplementation with Enriched Protein®: Participants will consume a low protein containing breakfast and 2 hours later will consume the enriched protein supplement
  Interventions: Dietary Supplement: Enriched Protein®
- Low protein breakfast: No supplementation
- High protein breakfast: No supplementation

INTERVENTIONS:
Dietary Supplement: Enriched Protein® — This product contains high quality bovine milk proteins enriched with additional leucine.
  Groups: Supplementation with Enriched Protein®

SUMMARY:
It is well known that dietary protein is a powerful transient stimulator of the muscle protein synthetic rate (MPS) whereby changes in MPS in response to feeding may be regulated by specific downstream target proteins of mammalian target of rapamycin signaling, such as S6K1, rpS6, and eIF2B. A meal deficient in protein, however, does not increase the rate of MPS because a rise in the bioavailability of amino acids does not occur. In addition, the source of dietary proteins has been shown to impact postprandial blood levels of amino acids. The concept that certain types of proteins are "fast acting" or "slow acting" has been shown to affect the postprandial profile of amino acids appearing in the systemic circulation. Native whey and micellar casein are both dairy proteins that contain a similar amount of essential (EAA), but blood EAA levels increase faster and to a higher level after the consumption of whey protein. Differences in gastric emptying, digestion and absorption kinetics between micellar casein and native whey are the underlying factors. Nonetheless, micellar casein protein has been shown to protract MPS in humans. Despite the significant amount of information gained with respect to both of these protein sources, the effects of combinatorial formulations on the postprandial profile of amino acids appearing in the blood is less well known. The purpose of the present study is to determine post-ingestion aminoacidemia, glycemia, and insulinemia from a specially formulated dairy protein blend.

DETAILED DESCRIPTION:
Experimental approach:

8 participants will be included in this study. Each participant will consume the supplement only once in a randomized fashion during three separate visits and there will be approximately 1 week between each visit.

Standardized meal:

Participants will be provided a standardized diet one day prior to experimentation. When performing research involving human metabolism it is important that the participants be tested in a weight-stable state. Therefore, the investigators will estimate the participants resting energy expenditure using a widely reference prediction formula, known as the Harris-Benedict equation. This formula takes into account gender, body mass, height, age, and self-reported activity level. Once resting energy expenditure is calculated the investigators will provide each participant with a pre-packaged standardized diet for the day prior to the experiment that is designed to ensure a sufficient energy balance.

Dual Energy X-Ray Absorptiometry (DXA) Scans:

DXA scans will be used to determine the participants body composition. The DXA procedures use a small amount of radiation to determine how much fat, bone, and lean mass the participants have in their body. The procedure takes approximately seven minutes and involves the participants lying still on an open bed while the sensor passes over the participants body.

Arterialized blood sampling:

All blood sampling will be achieved through an intravenous indwelling cannula. This method provides the least trauma to the participant when repeated blood sampling is required and is convenient for the investigators. In theory, repeated needle sticks may stress the participant thereby increasing sympathetic nervous system activity, thus causing changes in metabolism. Additionally, another potential drawback from venous blood sampling is the influence by regional tissue specific metabolism, thereby making it difficult to interpret whole-body metabolism on the basis of metabolites measured in venous blood. Therefore, arterial blood sampling is deemed the ideal method for metabolic studies. Arterial cannulation, however, may be unethical for research purposes due to increased risk of complications, such as damage to the arterial wall, thrombosis, and clot formation, all of which may cause death. Arterializing the blood being sampled can be achieved through heating either the superficial antecubital vein or dorsal hand vein with a heating blanket or specialized heat box. By doing so, blood flow increases as a result of vasodilatation of vessels in the arms skeletal musculature, as well as arteriovenous anastomoses in skin. Due to the increased blood flow and negligible muscle mass at the hand and elbow, results in venous blood being similar in composition to an arterial sample. This method is a widely used surrogate for safe direct arterial blood sampling. Once arterialized blood samples are obtained they will be preserved and used in analyses. The investigators will utilize heating blankets (Theratherm Large Digital Moist Heat Pad [14" x 27"]) to arterialize the blood samples and an infrared thermometer (Nubee, NUB8380) to determine the skin temperature (45-68∘C) prior to drawing the participant's blood.

Per-protocol conditions will include:

Consumption of a standardized meal the evening prior to each trial and consistent exercise/activity 2d before each trial There will be ~1wk between trials (washout periods) Blood samples will be analyzed for plasma amino acids, glucose, and insulin.

Experimental Interventions (randomized order):

1. Participants will consume a Low Protein Containing Breakfast (10% of the Acceptable Macronutrient Distribution Range according to the Food and Nutrition Board of the Institute of Medicine) and 2 hours later the participants will consume 17g of a leucine enriched whey protein- hydrolyzed whey protein-micellar casein blend (50:43:7 whey:hydrolyzed-whey:casein) containing 600 IU Vitamin D and 3.5g leucine
2. Participants will consume a High Protein Containing Breakfast (25% of the Acceptable Macronutrient Distribution Range according to the Food and Nutrition Board of the Institute of Medicine)
3. Participants will consume a Low Protein Containing Breakfast (10% of the Acceptable Macronutrient Distribution Range according to the Food and Nutrition Board of the Institute of Medicine)

Proteins were provided by Covance Laboratories, Inc. owned by Eurofins.

The whey protein and micellar casein are milk proteins derived from cow's milk. The participants will consume the 17g of protein contained in a semi-solid bar equal to ∼40g, which is the size of a typical sports recovery bar.

Sample size and data analyses:

The sample size was determined by a statistical power analysis (G*Power 3.1 software, version 3.1.9, 2014) that revealed a large effect size. This study was powered on the basis of previous studies. Thus, a total of 8 (n = 8/group) participants will be used in analyses. See Below:

Analysis: A priori: Compute required sample size ANOVA: Repeated measures, within-between interaction Input Effect size f = 0.5 α err prob = 0.05 Power (1-β err prob) = 0.95 Number of groups = 3 Number of measurements = 14 Corr. Among rep. measures = 0.5 Nonsphericity correction ε = 1 Output Noncentrality parameter ƛ = 63 Critical F = 1.6380186 Numerator df = 26 Denominator df = 78 Total sample = 9 Actual power = 0.997

ELIGIBILITY:
Inclusion Criteria:

* 8 participants will be included in this study. Each participant will consume the supplement only once in a randomized fashion during one of three separate visits and there will be approximately 1 week between each visit. In order to participate in this study, each participant must be male or female, 65 years or older (inclusive) and cannot be a smoker or user of tobacco products.

Exclusion Criteria:

* The exclusion requirements for this study include the following conditions:

  * Take any analgesic or anti-inflammatory drugs(s), prescription or non-prescription, chronically will be excluded. However, a washout period of 4 weeks will be suitable for participation.
  * A history of neuromuscular problems or muscle and/or bone wasting diseases
  * Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through medical history screening questionnaires
  * Use medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications)

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Healthy Older Adults
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Easy-fast amino acid sample testing kit for gas chromatography mass spectrometry | 375 minutes
  plasma amino acid concentrations

SECONDARY OUTCOMES:
Hexokinase/G-6-PDH methodology | 375 minutes
  plasma glucose concentrations
Chemiluminescent Microparticle Immunoassay | 375 minutes
  plasma insulin concentrations
Visual Analog Scale Questionnaires for food sensory perception desire to eat | Average score across 13 measurements
  Units on a 100mm Paper Scale, 0mm = lowest score and 100mm = highest score
Visual Analog Scale Questionnaires for food sensory perception for hunger | Average score across 13 measurements
  Units on a 100mm Paper Scale, 0mm = lowest score and 100mm = highest score
Visual Analog Scale Questionnaires for food sensory perception for fullness | Average score across 13 measurements
  Units on a 100mm Paper Scale, 0mm = lowest score and 100mm = highest score
Visual Analog Scale Questionnaires for food sensory perception for thirst | Average score across 13 measurements
  Units on a 100mm Paper Scale, 0mm = lowest score and 100mm = highest score
Visual Analog Scale Questionnaires for food sensory perception for how much food could be eaten | Average score across 13 measurements
  Units on a 100mm Paper Scale, 0mm = lowest score and 100mm = highest score
Visual Analog Scale Questionnaires for food sensory perception for liking or disliking of food | Average score across 13 measurements
  Units on a 100mm Paper Scale, 0mm = worst score and 100mm = best score
Visual Analog Scale Questionnaires for food sensory perception for visual appeal | Average score across 2 measurements
  Units on a 100mm Paper Scale, 0mm = worst score and 100mm = best score
Visual Analog Scale Questionnaires for food sensory perception for smell | Average score across 2 measurements
  Units on a 100mm Paper Scale, 0mm = worst score and 100mm = best score
Visual Analog Scale Questionnaires for food sensory perception for taste | Average score across 2 measurements
  Units on a 100mm Paper Scale, 0mm = worst score and 100mm = best score
Visual Analog Scale Questionnaires for food sensory perception for aftertaste | Average score across 2 measurements
  Units on a 100mm Paper Scale, 0mm = worst score and 100mm = best score
Visual Analog Scale Questionnaires for food sensory perception for pleasantness | Average score across 2 measurements
  Units on a 100mm Paper Scale, 0mm = worst score and 100mm = best score
Height in meters | One measurement at baseline
  Stadiometer
Weight in kilograms | One measurement at baseline
  Physician scale

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koopman R, Crombach N, Gijsen AP, Walrand S, Fauquant J, Kies AK, Lemosquet S, Saris WH, Boirie Y, van Loon LJ. Ingestion of a protein hydrolysate is accompanied by an accelerated in vivo digestion and absorption rate when compared with its intact protein. Am J Clin Nutr. 2009 Jul;90(1):106-15. doi: 10.3945/ajcn.2009.27474. Epub 2009 May 27. PMID 19474134
- [Result] Koopman R, Walrand S, Beelen M, Gijsen AP, Kies AK, Boirie Y, Saris WH, van Loon LJ. Dietary protein digestion and absorption rates and the subsequent postprandial muscle protein synthetic response do not differ between young and elderly men. J Nutr. 2009 Sep;139(9):1707-13. doi: 10.3945/jn.109.109173. Epub 2009 Jul 22. PMID 19625697
- [Result] Moore DR, Robinson MJ, Fry JL, Tang JE, Glover EI, Wilkinson SB, Prior T, Tarnopolsky MA, Phillips SM. Ingested protein dose response of muscle and albumin protein synthesis after resistance exercise in young men. Am J Clin Nutr. 2009 Jan;89(1):161-8. doi: 10.3945/ajcn.2008.26401. Epub 2008 Dec 3. PMID 19056590
- [Result] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. A high proportion of leucine is required for optimal stimulation of the rate of muscle protein synthesis by essential amino acids in the elderly. Am J Physiol Endocrinol Metab. 2006 Aug;291(2):E381-7. doi: 10.1152/ajpendo.00488.2005. Epub 2006 Feb 28. PMID 16507602
- [Result] Luiking YC, Abrahamse E, Ludwig T, Boirie Y, Verlaan S. Protein type and caloric density of protein supplements modulate postprandial amino acid profile through changes in gastrointestinal behaviour: A randomized trial. Clin Nutr. 2016 Feb;35(1):48-58. doi: 10.1016/j.clnu.2015.02.013. Epub 2015 Mar 5. PMID 25790724
- [Result] Tipton KD, Elliott TA, Cree MG, Wolf SE, Sanford AP, Wolfe RR. Ingestion of casein and whey proteins result in muscle anabolism after resistance exercise. Med Sci Sports Exerc. 2004 Dec;36(12):2073-81. doi: 10.1249/01.mss.0000147582.99810.c5. PMID 15570142
- [Result] Boirie Y, Dangin M, Gachon P, Vasson MP, Maubois JL, Beaufrere B. Slow and fast dietary proteins differently modulate postprandial protein accretion. Proc Natl Acad Sci U S A. 1997 Dec 23;94(26):14930-5. doi: 10.1073/pnas.94.26.14930. PMID 9405716
- [Result] Douglas CC, Lawrence JC, Bush NC, Oster RA, Gower BA, Darnell BE. Ability of the Harris Benedict formula to predict energy requirements differs with weight history and ethnicity. Nutr Res. 2007 Apr;27(4):194-199. doi: 10.1016/j.nutres.2007.01.016. PMID 19081830
- [Result] Churchward-Venne TA, Burd NA, Mitchell CJ, West DW, Philp A, Marcotte GR, Baker SK, Baar K, Phillips SM. Supplementation of a suboptimal protein dose with leucine or essential amino acids: effects on myofibrillar protein synthesis at rest and following resistance exercise in men. J Physiol. 2012 Jun 1;590(11):2751-65. doi: 10.1113/jphysiol.2012.228833. Epub 2012 Mar 25. PMID 22451437
- [Result] Churchward-Venne TA, Breen L, Di Donato DM, Hector AJ, Mitchell CJ, Moore DR, Stellingwerff T, Breuille D, Offord EA, Baker SK, Phillips SM. Leucine supplementation of a low-protein mixed macronutrient beverage enhances myofibrillar protein synthesis in young men: a double-blind, randomized trial. Am J Clin Nutr. 2014 Feb;99(2):276-86. doi: 10.3945/ajcn.113.068775. Epub 2013 Nov 27. PMID 24284442
- [Result] Copeland KC, Kenney FA, Nair KS. Heated dorsal hand vein sampling for metabolic studies: a reappraisal. Am J Physiol. 1992 Nov;263(5):E1010-4. doi: 10.1152/ajpendo.1992.263.5.E1010. PMID 1443110
- [Result] Green JH, Ellis FR, Shallcross TM, Bramley PN. Invalidity of hand heating as a method to arterialize venous blood. Clin Chem. 1990 May;36(5):719-22. PMID 2337978
- [Result] Tang JE, Moore DR, Kujbida GW, Tarnopolsky MA, Phillips SM. Ingestion of whey hydrolysate, casein, or soy protein isolate: effects on mixed muscle protein synthesis at rest and following resistance exercise in young men. J Appl Physiol (1985). 2009 Sep;107(3):987-92. doi: 10.1152/japplphysiol.00076.2009. Epub 2009 Jul 9. PMID 19589961
- [Result] Burd NA, West DW, Staples AW, Atherton PJ, Baker JM, Moore DR, Holwerda AM, Parise G, Rennie MJ, Baker SK, Phillips SM. Low-load high volume resistance exercise stimulates muscle protein synthesis more than high-load low volume resistance exercise in young men. PLoS One. 2010 Aug 9;5(8):e12033. doi: 10.1371/journal.pone.0012033. PMID 20711498
- [Derived] Traylor DA, Kamal M, Nunes EA, Prior T, Gorissen SHM, Lees M, Gesel F, Lim C, Phillips SM. Consumption of High-Leucine-Containing Protein Bar Following Breakfast Impacts Aminoacidemia and Subjective Appetite in Older Persons. Curr Dev Nutr. 2021 May 8;5(6):nzab080. doi: 10.1093/cdn/nzab080. eCollection 2021 Jun. PMID 34104852